CLINICAL TRIAL: NCT02734797
Title: Clinical Outcomes, Nutritional Status, Exercise and Psychosocial Factors in Pediatric Hematopoietic Cell Transplant
Acronym: CONSEPT
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2015.108; HUM00102331 (Other: The University of Michigan)
Record Dates: First submitted 2016-03-17; First posted 2016-04-12 (Estimated); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Malnutrition; Obesity
MeSH Terms: conditions — Malnutrition; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric patients: This is an observational study. Validated measures of nutritional status, dietary intake, body composition, functional status and psychosocial factors will be used to measure outcomes in study patients at 4 time-points: (1) pre-HCT (Baseline), (2) 30-days post-HCT, (3) 100-days post-HCT and (4) one year post-HCT.

SUMMARY:
Children who receive hematopoietic cell transplants (HCT) are at high nutritional risk due to comorbidities and complications that are likely to develop before, during and after transplant. Prior to transplant, many children undergo multiple rounds of chemotherapy which affect appetite and cause gastrointestinal toxicities that limit food intake. During transplant, painful mucositis makes it difficult to consume adequate nutrients and often children will require nutrition support such as parenteral or enteral nutrition. Energy imbalance and physical deconditioning following transplant can result in loss of lean body mass and functional impairment; these nutritional side effects are exacerbated if the child develops graft-versus-host disease. After transplant, a substantial number of childhood cancer survivors become overweight and develop metabolic syndrome. However, little is known about the prevalence and distribution of pediatric malnutrition (under-nutrition as well as obesity), the psychosocial factors that affect dietary intake and how the quality of the child's food intake and physical activity level throughout the transplant process might affect body composition and clinical outcomes. In this exploratory study, we will monitor nutritional status in pediatric patients undergoing HCT. This study will test the feasibility of collecting patient-reported dietary intake data along with anthropometric, body composition, functional status and psychosocial measurements that may influence dietary intake in pediatric patients undergoing HCT. The data collected in this preliminary analysis will inform future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric hematopoietic cell transplant patients, aged 2-25 years.
* Participants and/or at least one caregiver must speak, read and understand English.

Exclusion Criteria:

* Children younger than 2 years old at the time of their transplant or any child who is still breastfeeding will not be eligible due to the nature of the questionnaires and measurements.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric hematopoietic cell transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of comprehensive nutrition assessments in pediatric HCT patients | 1 year post-HCT
  Feasibility is defined as completion of comprehensive nutrition assessment by at least 50% of participants.

SECONDARY OUTCOMES:
Dietary intake | baseline (pre-HCT); day 30, day 100 and 1 year post-HCT
Determination of lean body mass measured using air displacement plethysmography (BOD POD) | baseline (pre-HCT); day 100 and 1 year post-HCT
Hand grip strength | baseline (pre-HCT); day 30, day 100 and 1 year post-HCT
PedsQL Pediatric Quality of Life Inventory | baseline (pre-HCT); day 30, day 100 and 1 year post-HCT
  Participants 10 years or older
PedsQL Cognitive Functioning Scale | baseline (pre-HCT); day 30, day 100 and 1 year post-HCT
  Participants 10 years or older
Dietary Patient Self-Efficacy Survey | baseline (pre-HCT); day 30, day 100 and 1 year post-HCT
  Participants 10 years or older

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No